CLINICAL TRIAL: NCT04921137
Title: A Randomised, Multicentre Trial Evaluating Harms and Benefits of Endocrine Therapy in Patients ≥70 Years of Age With Lower Risk Breast Cancer (REaCT-70)
Brief Title: Evaluating Harms and Benefits of Endocrine Therapy in Patients ≥70 Years of Age With Lower Risk Breast Cancer
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REaCT-70
Record Dates: First submitted 2021-05-27; First posted 2021-06-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Radiation therapy; Endocrine therapy; Older patients; Adjuvant therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omission of endocrine therapy (Experimental): Omission of endocrine therapy
  Interventions: Other: No endocrine therapy
- Administration of endocrine therapy for at least 5 years (Active Comparator): Administration of endocrine therapy for at least 5 years
  Interventions: Other: Endocrine therapy

INTERVENTIONS:
Other: No endocrine therapy — No endocrine therapy given
  Arms: Omission of endocrine therapy
Other: Endocrine therapy — Endocrine therapy given for at least 5 years
  Arms: Administration of endocrine therapy for at least 5 years

SUMMARY:
The current standard of care for stage 1 hormone receptor-positive (HR+) breast cancer consists of breast-conserving surgery followed by adjuvant radiotherapy (RT) and endocrine therapy (ET) for at least 5 years. The benefit of adjuvant ET for older patients is mitigated because of their increase risk of death from other causes and shorter time horizon to live. Clinical and pathological factors such as low-intermediate grade, tumor size ≤2 cm, and older age have been used in a few studies to identify patients with a lower risk of recurrence that might benefit from adjuvant therapy de-escalation, i.e. omission of RT or ET. Since there is no dedicated randomized clinical trial (RCT) conducted to evaluate the omission of ET, there is clinical equipoise as to whether we can omit adjuvant ET in older patients with lower-risk early-stage breast cancer. Therefore, we propose a randomised, multicentre trial evaluating harms and benefits of endocrine therapy in patients ≥70 years of age with lower risk breast cancer.

DETAILED DESCRIPTION:
The current standard of care for stage 1 hormone receptor-positive (HR+) breast cancer consists of breast-conserving surgery followed by adjuvant radiotherapy (RT) and endocrine therapy (ET) for at least 5 years. The benefit of adjuvant ET for older patients is mitigated because of their increase risk of death from other causes and shorter time horizon to live. This population is also more likely to have additional comorbidities which can lead to higher treatment-related adverse events impacting quality of life and precipitating functional decline. Clinical and pathological factors such as low-intermediate grade, tumor size ≤2 cm, and older age have been used in a few studies to identify patients with a lower risk of recurrence that might benefit from adjuvant therapy de-escalation, i.e. omission of RT or ET. The body of evidence from small prospective studies, mathematical modelling study and retrospective analyses would suggest that the omission of ET in older patients with favourable HR+ breast cancer who had optimal local therapy (i.e. breast conserving surgery followed by adjuvant radiotherapy) does not compromise locoregional and survival outcomes. Since there is no dedicated randomized clinical trial (RCT) conducted to evaluate the omission of ET, there is clinical equipoise as to whether we can omit adjuvant ET in older patients with lower-risk early-stage breast cancer. Therefore, we propose a randomised, multicentre trial evaluating harms and benefits of endocrine therapy in patients ≥70 years of age with lower risk breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* New invasive estrogen and/or progesterone receptor-positive (ER+ and/or PR+), HER2-negative (HER2-) invasive breast carcinoma diagnosis as per ASCO-CAP guidelines
* The primary tumour characteristics are either: Grade 1 and ≤5 cm on microscope exam, OR Grade 2 and ≤3 cm on microscope exam, OR Grade 3 and ≤1 cm on microscope exam
* Treated with standard loco-regional therapy: breast conserving surgery followed by adjuvant radiotherapy OR total mastectomy
* Axillary lymph node-negative (N0)
* Able to provide oral consent and complete questionnaires in French or English as per study protocol

Exclusion Criteria:

* Metastatic cancer

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Accrual of 100 participants across 8 centres within 2 years | 2 years after study initiation
  The accrual of at least 100 participants at 8 centres within 2 years.
Participation rate of at least 60% | 2 years after study initiation
  A participation rate of at least 60% among participants approached.
90% treatment allocation rate | 4 weeks after study enrolment
  At least 90% of enrolled participants receive treatment as per their allocated intervention for at least 4 weeks

SECONDARY OUTCOMES:
Significant adverse events | Baseline, 12 weeks, 26 weeks, 1 year, 2 years, 3 years, 4 years and 5 years after study enrolment
  Significant adverse events (e.g. bone fracture, stroke/transient ischemic attack, thromboembolic event, cardiac event, second cancer, hospitalization and death)
Endocrine therapy related toxicity | Baseline, 12 weeks, 26 weeks, 1 year, 2 years, 3 years, 4 years and 5 years after study enrolment
  Endocrine therapy (ET) related toxicity based upon Common Terminology for Adverse Events version 5 (CTCAEv5)
Health-related quality of life scores | Baseline, 12 weeks, 26 weeks, 1 year, 2 years, 3 years, 4 years and 5 years after study enrolment
  Health-related quality of life (HR-QoL) scores measured by the Cancer and Aging Research Group geriatric assessment (patient-tool) and the Functional Assessment of Cancer Therapy - Endocrine Symptom Subscale (FACT-B plus ES). The Cancer and Aging Research Group geriatric assessment tool (patient-tool) is utilized to capture information about a patient's medical history as well as functional, cognitive and psychosocial status. The FACT-B plus ES is used to measure the side effects and putative benefits of hormonal treatment given in breast cancer.
Rate of treatment discontinuation | 5 years after study enrolment
  The rate of endocrine therapy treatment discontinuations and reasons why the endocrine therapy treatment was discontinued.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Savard, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (7):
- Canada (7):
  - Grand River Hospital, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Oak Valley Health, Markham, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Savard MF, Clemons M, Hutton B, Jemaan Alzahrani M, Caudrelier JM, Vandermeer L, Liu M, Saunders D, Sienkiewicz M, Stober C, Cole K, Shorr R, Arnaout A, Chang L. De-escalating adjuvant therapies in older patients with lower risk estrogen receptor-positive breast cancer treated with breast-conserving surgery: A systematic review and meta-analysis. Cancer Treat Rev. 2021 Sep;99:102254. doi: 10.1016/j.ctrv.2021.102254. Epub 2021 Jun 19. PMID 34242928
- [Background] Alzahrani M, Clemons M, Chang L, Vendermeer L, Arnaout A, Larocque G, Cole K, Hsu T, Saunders D, Savard MF. Management Strategies for Older Patients with Low-Risk Early-Stage Breast Cancer: A Physician Survey. Curr Oncol. 2021 Dec 21;29(1):1-13. doi: 10.3390/curroncol29010001. PMID 35049675
- [Background] Savard MF, Alzahrani MJ, Saunders D, Chang L, Arnaout A, Ng TL, Brackstone M, Vandermeer L, Hsu T, Awan AA, Cole K, Larocque G, Clemons M. Experiences and Perceptions of Older Adults with Lower-Risk Hormone Receptor-Positive Breast Cancer about Adjuvant Radiotherapy and Endocrine Therapy: A Patient Survey. Curr Oncol. 2021 Dec 8;28(6):5215-5226. doi: 10.3390/curroncol28060436. PMID 34940075
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/